CLINICAL TRIAL: NCT03634813
Title: Perioperative Blood Pressure Screening to Improve Long-term Cardiovascular Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2000023093
Record Dates: First submitted 2018-08-10; First posted 2018-08-16 (Actual); Results first posted 2021-05-24 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Blood Pressure

STUDY DESIGN:
Intervention Model Description: 2 cohort parallel
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- High Blood Pressure Monitoring and Counseling (Experimental): Enrolled patients will be fitted with a HBPM device and instructed in its use. Patients will be asked to return the HBPM device on the morning of surgery. At the same time they receive the HBPM device, they will also be provided with the National Institutes of Health (NIH) booklet called "Your guide on lowering blood pressure", which has several guidelines regarding diet, exercise and lifestyle changes that can be implemented to improve blood pressure control.
  Interventions: Device: High Blood Pressure Monitor
- Usual Care (Active Comparator): The usual care group will receive brief counseling after the PAT visit which will review their blood pressure readings taken at the clinic and how they compare with the American Heart Association (AHA) blood pressure guidelines. They will be offered the suggestion that they should follow up with their primary care doctor 2-4 weeks after their surgical episode is completed, or at their earliest convenience.
  Interventions: Procedure: Usual Care

INTERVENTIONS:
Device: High Blood Pressure Monitor — High Blood Pressure Monitoring device (Omron MX3 model BP742, Omron, Shaumberg, IL)
  Arms: High Blood Pressure Monitoring and Counseling
Procedure: Usual Care — Usual Care
  Arms: Usual Care

SUMMARY:
To explore in a pilot randomized clinical trial, the impact of Home Blood Pressure Monitoring with patient directed information as compared to usual care on the postoperative management of blood pressure.

DETAILED DESCRIPTION:
The intervention and control groups will be defined by, 1) preoperative home blood pressure monitoring with a detailed report sent to the patient, and 2) usual standard of care including a suggestion during the pre-operative clinic appointment to follow up with Primary Care. Both groups will receive a brief questionnaire about their blood pressure treatment and medication adherence. We will examine the rate of primary care follow-up and changes in hypertension treatment at 60 days post-operative, through a telephone call. This information, along with information regarding patient acceptance of the intervention will be used to inform the design of a future clinical trial powered to outcomes, including follow-up visits and blood pressure management.

ELIGIBILITY:
Inclusion Criteria:

* We propose to recruit patients who present for ambulatory surgery, aged >18 years, with a preoperative blood pressure > 140/90 mmHg taken as the mean of two readings during the pre-admission testing visit.

Exclusion Criteria:

* Patients who are unable or unwilling to be contacted by telephone, are non-English speaking, or are unable to operate an automated home blood pressure monitor will also be excluded.
* Healthy patients with blood pressure readings that fall within the American Heart Association (AHA) guidelines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-08-31 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2021-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Schonberger, MD, Principal Investigator — Yale University
Locations (1):
- Yale-New Haven Hospital PreAdmission Testing Clinic, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Diaz SI, Yan L, Dai F, Zhou B, Burg MM, Schonberger RB. Feasibility of a randomized hypertension screening initiative in the perioperative setting. Perioper Med (Lond). 2021 Nov 22;10(1):39. doi: 10.1186/s13741-021-00210-7. PMID 34802471

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High Blood Pressure Monitoring and Counseling | Usual Care
Started | 49 | 51
Completed | 49 | 51
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Usual Care: The usual care group will receive brief counseling after the PAT visit which will review their blood pressure readings taken at the clinic and how they compare with the American Heart Association (AHA) blood pressure guidelines. They will be offered the National Institutes of Health (NIH) booklet called "Your guide on lowering blood pressure". They will be offered the suggestion that they should follow up with their primary care doctor 2-4 weeks after their surgical episode is completed, or at their earliest convenience.
  Usual Care: Usual Care
- Total: Total of all reporting groups
Arm/Group | High Blood Pressure Monitoring and Counseling | Usual Care | Total
Number analyzed (Participants) | 49 | 51 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (13.5) | 64.5 (9.6) | 64.9 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 27 | 54
  Male | 22 | 24 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 9 | 20
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 38 | 42 | 80
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 11 | 16
  White | 39 | 33 | 72
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Patients Reporting Primary Care Follow-up
Description: For the primary analysis, we will estimate the proportion of subjects that had a primary care follow-up visit within 60 days
Time Frame: 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | High Blood Pressure Monitoring and Counseling | Usual Care
Number analyzed (Participants) | 49 | 51
Participants | 36 | 36

2. Primary Outcome: Patients Reporting New/Adjusted Hypertension Treatment.
Description: For the primary analysis, we will estimate the proportion reporting new/adjusted hypertension treatment within 60 days. The count of participants is the number of patients for whom it was determined that they had new or adjusted hypertension treatment.
Time Frame: 60 days
Population: The overall number of participants analyzed were those successfully reached or whose ehr information enabled determination of the outcome in each arm.
Measure: Count of Participants; unit: Participants
Groups:
- Usual Care: The usual care group will receive brief counseling after the PAT visit which will review their blood pressure readings taken at the clinic and how they compare with the American Heart Association (AHA) blood pressure guidelines; they will also be provided with the National Institutes of Health (NIH) booklet called "Your guide on lowering blood pressure". They will be offered the suggestion that they should follow up with their primary care doctor 2-4 weeks after their surgical episode is completed, or at their earliest convenience.
  Usual Care: Usual Care
Arm/Group | High Blood Pressure Monitoring and Counseling | Usual Care
Number analyzed (Participants) | 31 | 36
Participants | 18 | 17

3. Secondary Outcome: Patient Acceptance/Satisfaction With Blood Pressure Care
Description: Patient Acceptance/Satisfaction With Blood Pressure Care. A questionnaire was provided to all participants, these data were not intended to be compared between treatment arms. The count of participants is the number of participants that reported they were moderately to very satisfied with their care.
Time Frame: 60 days
Population: 61 total patients that completed the questionnaire.
Measure: Count of Participants; unit: Participants
Arm/Group | High Blood Pressure Monitoring and Counseling | Usual Care
Number analyzed (Participants) | 31 | 30
Participants | 26 | 26

4. Other Pre Specified Outcome: Patients Demonstrating HBPM Elevation.
Description: The proportion of patients demonstrating HBPM elevation was measured. Specific cut-offs for the interpretation of home blood pressure are controversial. The mean home blood pressure threshold was > 135/85 mmHg as indicating hypertension, in-line with recommendations from the American Heart Association.
Time Frame: 1 year
Population: 3 of the devices were not returned.
Measure: Count of Participants; unit: Participants
Groups:
- HBPM Group Only: HBPM participants only
Arm/Group | HBPM Group Only
Number analyzed (Participants) | 46
Participants | 36

ADVERSE EVENTS:
Time Frame: 60 days
Arm/Group | High Blood Pressure Monitoring and Counseling | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/51
Other Adverse Events (participants affected / at risk) | 0/49 | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-16): https://cdn.clinicaltrials.gov/large-docs/13/NCT03634813/Prot_SAP_001.pdf